CLINICAL TRIAL: NCT04778566
Title: Evaluating the Cologuard Test for Use in Lynch Syndrome
Status: Withdrawn | Type: Observational
Why Stopped: Recent discovery of a novel assay that is more likely to be beneficial for patients with Lynch Syndrome. Investing into current version of Cologuard test would provide little clinical benefit.
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Rajiv Panikkar, Sponsor - Investigator, Geisinger Clinic
Other Study IDs: 2020-0239
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Lynch Syndrome; Colorectal Cancer; Colonic Adenoma; Colonic Polyp
Keywords: Lynch Syndrome; Colorectal Cancer; Hereditary non-polyposis colon cancer; High-Risk Colon Cancer; Health-Related Quality of Life; Bowel Prep Tolerability; Colonoscopy; Procedural anxiety
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Colorectal Neoplasms; Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cologuard Study Group: Within 60 days of their already scheduled screening colonoscopy, participants will provide a stool sample to be tested by a Cologuard screening test kit. Participants will also complete surveys prior to their colonoscopy as well as post colonoscopy.
  Interventions: Diagnostic Test: Cologuard test

INTERVENTIONS:
Diagnostic Test: Cologuard test — Cologuard is a stool-DNA screening test for detecting colon cancer

SUMMARY:
This study is aiming to enroll 90 patients with genetically confirmed Lynch Syndrome (LS) from Geisinger's High Risk Colorectal Cancer Clinic (HRC). Upon enrollment in the study, a Cologuard test will be ordered and the results will be blinded until data analysis. Patients enrolled in the study will also undergo a colonoscopy as part of their routine HRC visit.

DETAILED DESCRIPTION:
The primary aim is to perform a pilot study to gain information toward the implementation of a larger prospective study that will compare the performance of Cologuard with the gold-standard colonoscopy in identifying advanced adenomas and colorectal cancers in LS. Data regarding rate of consent, and adherence to the protocol will be recorded. Since patients with known genetic predisposition to cancers tend to view screening tests more positively than the general population, a second aim of the study is to evaluate patient satisfaction with bowel preparation, colonoscopies, and Cologuard testing. Up to 90 individuals with genetically confirmed LS will be recruited via Geisinger's HRC to complete a goal of 90 Cologuard studies. Upon enrollment, Cologuard will be ordered by the study team at no cost to the subject and will be completed according to the standard instructions for use. Results will be securely obtained and blinded until the time of data analysis. Subjects will undergo colonoscopy as part of their routine HRC visit. Results from the colonoscopy (and biopsy as indicated) will be retrieved from the Electronic Health Record (EHR) and documented in a research-associated spreadsheet. If repeat colonoscopy is clinically indicated, repeat Cologuard may be completed if the subject meets inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-89
* Diagnosis of genetically confirmed LS
* Scheduled for standard of care colonoscopy within 60 days of enrollment

Exclusion Criteria:

* Diagnosis of other inherited genetic disorders that increase risk for Colorectal Cancer (CRC) (Familial Adenomatous Polyposis (FAP), Cowden's syndrome, Turcot syndrome, Gardner syndrome, and Peutz-Jeghers syndrome)
* Diagnosis of other inherited Inflammatory bowel disease (i.e. Crohn disease, ulcerative colitis)
* Others with elevated risk of CRC outside of the inclusion criteria (i.e. ≥2 first-degree relatives who have been diagnosed with CRC without a defined inherited genetic disorder, Hereditary Non-Polyposis Colon Cancer (HNPCC) without genetic confirmation of LS)
* Participation in any interventional clinical study within the previous 30 days
* Personal history of CRC not in full remission (5 consecutive cancer-free years)
* Current active treatment with chemotherapy
* Treatment with chemotherapy within 12 months prior to consent date

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients being followed in the HRC with a diagnosis of LS
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the feasibility of the Cologuard test for Lynch Syndrome | 3 months
  To evaluate the feasibility of Cologuard in a high-risk population, a summary report of the enrollment/consent rate and adherence to the protocol will be provided. Additional analyses comparing the results (given as positive/negative) Cologuard with the gold standard of colonoscopy will be performed using diagnostic tests including sensitivity, specificity, positive predictive value and negative predictive value.

SECONDARY OUTCOMES:
Evaluate patient satisfaction with Cologuard | 3 months
  To evaluate patient satisfaction of Cologuard the responses to the Geisinger Cologuard Satisfaction Questionnaire will be summarized. The questionnaire is composed of 15 questions. There are two primary questions are "How satisfied are you with the process of using Cologuard which uses a 5 point Likert Scale (Very satisfied to Very Dissatisfied) and "would you recommend Cologuard using a 10 point Likert scale (Not at all likely to Extremely Likely). Other categorical questions are either yes no response or an ordinal response with 4 categories. There are 6 questions that are open text responses to give more details as to why the selected their categorical response. The information gathered in the open responses is qualitative and will be used to provide guidance of approach and protocol for a future study.
Evaluate health-related quality of life in Lynch Syndrome | 3 months
  Assess the results of the 12-Item Short Form Health Survey (SF-12) collected at the initial subject contact. Responses will be summarized.
Evaluate depressive symptoms | 3 months
  Assess the results of the Patient Health Questionnaire - 9 (PHQ-9) collected at the time of their High-Risk Clinic Visit. Responses will be summarized.
Evaluate anxiety symptoms surrounding routine colonoscopy | 3 months
  Assess the results of the General Anxiety Disorder - 7 item scale (GAD-7) collected at the initial subject contact and that collected at the completion of their participation. Responses will be summarized
Evaluate bowel preparation tolerability | 3 months
  Assess the results of the Mayo Florida Bowel Prep Tolerability Questionnaire (MFBT-9) collected at the completion of the subject's participation. Responses will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Panikkar, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No